CLINICAL TRIAL: NCT04172311
Title: Modified Atkins Diet Versus Levetiracetam for Refractory Epilepsy in Children: A Randomized Open-Label Study
Brief Title: Modified Atkins Diet Versus Levetiracetam for Refractory Childhood Epilepsy
Acronym: LEVEMAD
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, Suvasini Sharma, Associate Professor, Lady Hardinge Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEVEMAD
Record Dates: First submitted 2019-11-15; First posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Refractory Childhood Epilepsy
MeSH Terms: interventions — Levetiracetam

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Modified Atkins Diet (Experimental): Modified Atkins Diet administration
  1. Carbohydrates will be restricted to 10 grams per day.
  2. Recipes will be provided to be prepared from easy home available foods, to have 2.5 gram per meal. Along with this, a list of carbohydrate free foods will be provided.
  3. Fats intake will be actively encouraged. Protein intake will be unrestricted.
  4. Medications will be changed to carbohydrate free preparations.
  5. A multivitamin and calcium supplementation will be added.
  Interventions: Other: Modified Atkins Diet
- Levetiracetam (Active Comparator): Levetiracetam will be started at a dose of 10 mg/kg/day in two divided doses and increased to 20 mg/kg/day after 1 week. Syrups will be used in children younger than 5 years of age, and tablets will be used in children > 5 years of age. Further dose titration will be done as per the seizure control, in 10 mg/kg/day increments in 2 weekly intervals, to a maximum of 60mg/kg/day.
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Other: Modified Atkins Diet — Modified Atkins diet is a type of ketogenic diet which is less restrictive
  Other Names: Ketogenic Diet subtype
  Arms: Modified Atkins Diet
Drug: Levetiracetam — Levetiracetam is a second generation anti-epileptic drug which is broad spectrum and commonly used as add-on in refractory epilepsy
  Arms: Levetiracetam

SUMMARY:
In this study, the efficacy of add-on modified Atkins diet will be compared with add-on Levetiracetam in children with refractory epilepsy in a randomized open label trial. The results will aid clinicians in deciding the treatment options when a child has been diagnosed to have refractory epilepsy.

DETAILED DESCRIPTION:
Epilepsy is a disorder of the brain characterized by an enduring predisposition to generate seizures and by the neurobiologic, cognitive, psychological and social consequences of this condition. Epilepsy is a disabling and common neurological condition which rank 4th in the world's neurological disorder burden, which can be controlled successfully in most of the patients with one or more antiepileptic drugs. But approximately 30% of patients with epilepsy have refractory epilepsy, which is, a failure to respond to adequate trials of two tolerated, appropriately chosen and used antiepileptic drug schedules to achieve sustained relief of seizures.Many severe and catastrophic epilepsies present in children such as West syndrome, Lennox Gastaut syndrome, Dravet syndrome. Uncontrolled epilepsy carries significant risks for the affected child, such as injuries, cognitive and behavioural problems. Epilepsy surgery is a good option but it is expensive and not easily available. Also, many children with refractory epilepsy are not good surgical candidates. Hence there is a need to consider alternative treatments in these children.

The ketogenic diet is an individually calculated and rigidly controlled high-fat, low carbohydrate diet used for the treatment of difficult to control seizures. The ketogenic diet is an effective treatment option for refractory childhood epilepsy however it is very restrictive and difficult to implement in low resource settings. The modified Atkins diet is a less restrictive alternative to the traditional ketogenic diet. This diet is started on an outpatient basis without a fast, and allows unlimited protein and fat. This diet has been shown to be equally effective as the ketogenic diet and a useful option in resource-constraint settings. The modified Atkins diet has been demonstrated to be effective in refractory childhood epilepsy in two randomized controlled trials from India. However, in both these trials the control groups continued their ongoing antiepileptic medication without any new treatment.

Levetiracetam is one of the newer antiepileptic drugs available for treating drug resistant epilepsy. It is a broad-spectrum antiepileptic drug effective in most seizure types. It also has an excellent pharmacokinetics and tolerability profile with no known pharmacokinetic interactions. Use of levetiracetam as an add on drug in refractory childhood epilepsy recently in some published studies has shown good efficacy.

In this study, the efficacy of add-on modified Atkins diet will be compared with add-on Levetiracetam in children with refractory epilepsy in a randomized open label trial. The results will aid clinicians in deciding the treatment options when a child has been diagnosed to have refractory epilepsy.

ELIGIBILITY:
Inclusion Criteria:

Seizures persisting more than 3 per week despite the use of at least 2 appropriate anti-epileptic drugs in appropriate doses -

Exclusion Criteria:

1. Known or suspected inborn error of metabolism
2. Surgically remediable causes of epilepsy such as tumours, cortical dysplasia, mesial temporal lobe epilepsy etc with refractory focal epilepsy.
3. Prior use of the ketogenic or modified Atkins diet or levetiracetam.
4. Systemic illness- chronic hepatic, renal or pulmonary disease
5. Prior history of depression or severe behavioural problems.

   -

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2019-11-14 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-04-20 (Estimated)

PRIMARY OUTCOMES:
Efficacy in reducing seizures measured by The proportion of responders, i.e., patients who achieve > 50% seizure reduction from the baseline in the modified Atkins diet group at 3 months in comparison to the levetiracetam group. | 3 months
  The proportion of responders, i.e., patients who achieve > 50% seizure reduction from the baseline in the modified Atkins diet group at 3 months in comparison to the levetiracetam group.

SECONDARY OUTCOMES:
Treatment emergent adverse effects in both groups | 3 months
  Tolerability and the adverse effects of the modified Atkins diet and levetiracetam

CONTACTS AND LOCATIONS:
Locations (1):
- Lady Hardinge Medical College, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No